CLINICAL TRIAL: NCT00402558
Title: Alloreactive NK Cells With Busulfan, Fludarabine and Thymoglobulin for Allogeneic Stem Cell Transplantation for AML and MDS
Brief Title: Alloreactive NK Cells for Allogeneic Stem Cell Transplantation for Acute Myeloid Leukemia (AML) and Myelodysplastic Syndrome (MDS)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2005-0508; NCI-2012-01484 (Registry Identifier: NCI CTRP); 1P01CA100265 (NIH)
Record Dates: First submitted 2006-11-20; First posted 2006-11-22 (Estimated); Last update posted 2015-05-08 (Estimated); Status verified 2015-05

CONDITIONS: Myelodysplastic Syndrome; Leukemia
Keywords: Acute Myeloid Leukemia; Chronic Myelogenous Leukemia; Myelodysplastic Syndrome; Leukemia; NK Cells; Natural Killer Cells; Fludarabine; Busulfan; Thymoglobulin; AML; CML; MDS; ATG; Antithymocyte globulin; Busulfex; Myleran®; Fludarabine Phosphate; G-CSF; Filgrastim; Neupogen; Interleukin-2; IL-2; Aldesleukin; Proleukin; Tacrolimus; Prograf; Methotrexate
MeSH Terms: conditions — Myelodysplastic Syndromes; Leukemia; Leukemia, Myeloid, Acute; Leukemia, Myelogenous, Chronic, BCR-ABL Positive | interventions — thymoglobulin; Antilymphocyte Serum; Busulfan; fludarabine; fludarabine phosphate; Granulocyte Colony-Stimulating Factor; Filgrastim; Tacrolimus; Methotrexate; Interleukin-2; aldesleukin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Thymoglobulin + Busulfan + Fludarabine (Experimental): Thymoglobulin 1.5 mg/kg by vein for 3 days. Busulfan 130 mg/m^2 by vein for 4 days. Fludarabine 40 mg/m^2 by vein for 4 days. Alloreactive NK infusion from haploidentical donor on Day -8. Alloreactive NK cell infusion given at one of 4 dose levels 10e6, 5 x 10e6, 3 x 10e7 cells/kg and 3 x10e7 NK Cells plus systemic interleukin-2 treatment. The 4th dose level is 3 x 107 NK cells/kg plus systemic interleukin-2 at a dose of 0.5 million units per day subcutaneously starting on Day -8 (day of the NK cell infusion) to Day -4.
  G-CSF 5 mcg/kg/day subcutaneously beginning on Day +7, and continuing until absolute neutrophil count is > 500 x 109/L for 3 consecutive days. Tacrolimus starting dose of 0.015 mg/kg daily adjusted to achieve a therapeutic level of 5-15 ng/ml. Tacrolimus changed to oral dosing when tolerated and can be tapered off after Day +90 if no GVHD is present. Methotrexate 5 mg/m2 by vein on Days 1, 3 and 6 and Day +11 post transplant.
  Interventions: Drug: Thymoglobulin; Drug: Busulfan; Drug: Fludarabine; Procedure: Alloreactive NK Infusion; Drug: G-CSF; Drug: Tacrolimus; Drug: Methotrexate; Drug: Interleukin-2

INTERVENTIONS:
Drug: Thymoglobulin — 1.5 mg/kg By Vein Daily x 3 Days
  Other Names: ATG; Antithymocyte globulin
Drug: Busulfan — 130 mg/m^2 By Vein Over 3 Hours x 4 Days
  Other Names: Busulfex; Myleran®
Drug: Fludarabine — 40 mg/m^2 By Vein Over 30 Minutes x 4 Days
  Other Names: Fludarabine Phosphate; Fludara
Procedure: Alloreactive NK Infusion — Alloreactive NK infusion from haploidentical donor on Day -8. The alloreactive NK cell infusion given at one of 4 dose levels 10e6, 5 x 10e6, 3 x 10e7 cells/kg and 3 x10e7.
Drug: G-CSF — 5 mcg/kg/day subcutaneously beginning on Day +7, and continuing until absolute neutrophil count (ANC) is > 500 x 109/L for 3 consecutive days.
  Other Names: Filgrastim; Neupogen
Drug: Tacrolimus — Starting dose of 0.015 mg/kg as a 24 hour continuous infusion daily adjusted to achieve a therapeutic level of 5-15 ng/ml. Tacrolimus changed to oral dosing when tolerated and can be tapered off after Day +90 if no GVHD is present.
  Other Names: Prograf
Drug: Methotrexate — 5 mg/m2 intravenously on Days 1, 3 and 6 and Day +11 post transplant.
Drug: Interleukin-2 — 0.5 million units per day subcutaneously starting on Day -8 (day of the NK cell infusion) to Day -4 only to participants receiving fourth dose level of NK cells.
  Other Names: Aldesleukin; IL-2; Proleukin

SUMMARY:
The goal of this clinical research study is to determine the safety and effects of giving a special kind of immune cells called "alloreactive natural killer (NK) cells" with high dose chemotherapy and allogeneic hematopoeitic stem cell transplantation with the goal of defining the maximum tolerated dose of NK cells. The NK cells will be donated from a relative of yours who has certain genetic type in their blood called HLA, that almost matches yours. The stem cells you will receive will come from a separate HLA matched (HLA A, B, C, DR) relative or unrelated donor. The safety of this treatment will also be studied.

DETAILED DESCRIPTION:
NK cells are part of the immune system (the cells in your body that fight disease). Sometimes, NK cells react against and fight leukemia cells that are mismatched with your body for certain HLA tissue type proteins. When the NK cells react, these cells are called "alloreactive NK cells."

In this study, researchers will collect alloreactive NK cells from the blood of a relative of yours whose HLA proteins do not match yours exactly. The NK cells are separated from the blood using a machine called a CLINIMACs system. This machine uses special kinds of cells and magnetic beads to separate the NK cells. The drug interleukin-2 is then added to the NK cells, to improve their function. The interleukin-2 will be washed out of the cell sample before it is given to you. The CliniMACS System is a medical device that is used to separate types of blood cells from blood that is removed from the body during leukapheresis. These separated cells are processed for use in treatments such as stem cell transplants.

If you are able to take part in this study, you will receive high-dose chemotherapy for 4 days. You will receive fludarabine over about 30 minutes daily as an intravenous (IV--through a needle in your vein) infusion . You will also receive busulfan over 3 hours by IV once a day. About 2 days later, you will be given the infusion of the alloreactive NK cells by IV. Patients will receive one of 3 dose levels. Some patients will receive interleukin-2 daily for 4 days to enhance the function of the NK cells.

Five (5) days after the NK cell infusion, thymoglobulin will be given to you by IV daily for 3 days. Thymoglobulin is an immunosuppressive treatment to reduce the risk of graft rejection. Then blood stem cells will be administered IV from a different stem cell donor whose HLA type matches yours.

You will receive the drugs tacrolimus and methotrexate to help lower the risk of a reaction called "graft-vs.-host disease" (GVHD). GVHD is when the donated immune cells in the transplant react against the body of the person receiving the cells. Tacrolimus will be given by IV for about 2 weeks, and after that it is given by mouth as a pill for at least 3 months. Methotrexate will be given as an IV injection for 3 to 4 doses over the first 11 days after the stem cell transplant.

You will also receive the drug G-CSF (Neupogen) as an injection under the skin until your blood cell counts reach a certain high enough level.

You will need to stay in the hospital for about 4 weeks. After you leave the hospital, you will continue as an outpatient in the hospital area, which means you will have to stay close enough to be able to come back for any visits for at least 100 days after the transplant.

You will be asked to come back to the clinic at 3, 6, and 12 months after your transplant for routine safety testing. This will include a physical exam, a bone marrow biopsy, and routine blood draws.

This is an investigational study. The way the researchers make the alloreactive NK cells using the CLINIMACs device is investigational. The CliniMACS device is not FDA approved. At this time, it is being used in research only. Up to 18 patients will take part in this study.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with age </= 70 years with one of of the following: Acute myeloid leukemia past first remission, in first or subsequent relapse, in second or greater remission or primary induction failure; Myelodysplastic syndromes with intermediate or high risk IPSS score; CML which has progressed to accelerated phase or blast crisis despite imatinib treatment
2. Patients must have an HLA matched (HLA A, B, C, DR) related or unrelated donor willing to donate for allogeneic peripheral blood progenitor cell transplantation. (Recent large analyses of the National Marrow Donor Program indicate that a mis-match at the DQ locus has no adverse effect on outcome. The current national standard of care is to consider only these 4 loci in identifying suitably "matched" donors.)
3. Patients must have a haploidentical relative who is predicted to be alloreactive based upon the presence of the relevant KIR genes and incompatibility with the recipient for HLA C and Bw antigens.
4. Zubrod performance status </= 2.
5. Left ventricular ejection fraction >/= 45%. No uncontrolled arrhythmias or uncontrolled symptomatic cardiac disease.
6. No symptomatic pulmonary disease. forced expiratory volume at one second (FEV1), forced vital capacity (FVC) and diffusing capacity of lung for carbon monoxide (DLCO) >/= 50% of expected, corrected for hemoglobin.
7. Serum creatinine </= 1.8mg%.
8. Serum glutamate pyruvate transaminase (SGPT) </= 200 IU/ml unless related to patients malignancy.
9. Bilirubin </= 1.5 mg/dl (unless Gilbert's syndrome).No evidence of chronic active hepatitis or cirrhosis. If positive hepatitis serology, discuss with Study Chairman and consider liver biopsy.
10. Patient or patient's legal representative, parent(s) or guardian able to sign informed consent.
11. No known allergy to mouse proteins or monoclonal antibodies

Exclusion Criteria:

1. Uncontrolled infection, not responding to appropriate antimicrobial agents after seven days of therapy. The Protocol PI is the final arbiter of eligibility.
2. Pleural/pericardial effusion or ascites estimated to be >1L.
3. HIV-positive.
4. Pregnancy: Positive Beta Human Chorionic Gonadotropin (HCG) test in a woman with child bearing potential defined as not post-menopausal for 12 months or no previous surgical sterilization.
5. Known allergy to mouse proteins.
6. Patient has received other systemic chemotherapeutic drugs (including Mylotarg) within 14 days prior to trial enrollment or has unresolved grade >1 toxicity from prior chemotherapy treatment. (Hydroxyurea or low dose ara-c less than or equal to 20 mg/m2/d is permitted if indicated to control induction refractory disease, and IT chemotherapy is allowed if indicated as maintenance treatment for previously diagnosed lumbar microdiscectomy (LMD), that is in remission prior to enrollment on this study).

Max Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2006-05; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose of NK cells | Continual Reassessment (Baseline, 3, 6 and 12 Months Follow Ups)

CONTACTS AND LOCATIONS:
Overall Officials: Richard E. Champlin, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org